CLINICAL TRIAL: NCT04282473
Title: Peristomal Hernia Rate 5 Years After a Terminal Colostomy With the Parietex ™ TCM Parietal Prosthesis Versus Without Mesh: Material-epidemiology Study
Brief Title: Peristomal Hernia Rate 5 Years After a Terminal Colostomy With the Parietex ™ TCM Parietal Prosthesis Versus Without Mesh
Acronym: RESEDAE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2018-02/MP-01
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Colostomy Stoma; Parastomal Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with mesh: Placement of lightweight (<50g/m2) monofilament mesh during colostomy formation
- no mesh: colostomy without mesh placement

SUMMARY:
This study is a follow-up of the GRECCAR 07 cohort (NCT01380860). Patients will be evaluated 5 years following terminal colostomy to observe patient long-term patient outcomes from colostomy with and without mesh placement.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be affiliated with a health insurance programme
* Patient was included in the GRECCAR 07 cohort (PHRC National 2011; N° RCB: 2011-A01572-39 - ClinicalTrials.gov ID: NCT01380860)
* Patient received colostomy 5 years ago

Exclusion Criteria:

* The subject is participating in another category I interventional study, or is in a period of exclusion determined by a previous study
* The subject signals opposition to participating in the study
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients included in the GRECCAR 07 cohort.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of parastomal hernia between groups | 5 years after colostomy formation
  Percentage patients with parastomal hernia taken from patient medical records
Date of parastomal hernia | 5 years after colostomy formation
  Date of parastomal hernia taken from patient records

SECONDARY OUTCOMES:
Protrusion around the stoma | 5 years after colostomy formation
  Yes/no
Patient reported pain | 5 years after colostomy formation
  Yes/no
Occlusion | 5 years after colostomy formation
  Yes/no
Incarceration | 5 years after colostomy formation
  Yes/no
Patient reported quality of life | 5 years after colostomy formation
  Stoma-QoL questionnaire - a 20-item questionnaire on a four-point Likert scale with total score ranging from 0 (worst score) to 100 (best score)
Pain at colostomy site | 5 years after colostomy formation
  0-100 scale (no pain to intolerable pain)
Discomfort | 5 years after colostomy formation
  0-100 scale (very uncomfortable to very comfortable)
Patient reported satisfaction | 5 years after colostomy formation
  0-100 scale (not at all satisfied to very satisfied)
Number of specialist and general consultations attended by patients between groups | 5 years after colostomy formation
  number of consultations
Number of medications taken in each group | 5 years after colostomy formation
  Number of medications taken
Other associated treatment received by patients in each group | 5 years after colostomy formation
  number of treatments received
Rehabilitation sessions undergone by patients in each group | 5 years after colostomy formation
  number of rehabilitation sessions
Sick leave taken by patients in each group | 5 years after colostomy formation
  Number of days
Cost of patients care | 5 years after colostomy formation
  Euros

CONTACTS AND LOCATIONS:
Overall Officials: Michel Prudhomme, MD, Principal Investigator — CHU Nimes
Locations (16):
- France (16):
  - L'Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHRU Clermont- Ferrand Hôtel -Dieu, Clermont-Ferrand
  - Hôpital Beaujon (AP-HP), Clichy
  - Hôpital Albert Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Lyon-Sud, Lyon
  - Centre Régional de Lutte contre le Cancer Institut Paoli-Calmettes, Marseille
  - Hôpital La Timone, AP-HM, Marseille
  - CRLC Val d'Aurelle - Paul Lamarque, Montpellier
  - Centre Hospitalier Universitaire Hôtel-Dieu - CHU de Nantes, Nantes
  - CHU de Nimes, Nîmes
  - Hôpital Saint Antoine (AP-HP), Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles-Nicolle, Rouen
  - Hôpital Purpan - CHU de Toulouse, Toulouse